CLINICAL TRIAL: NCT07084428
Title: Pancreatic Antibiotic Concentration Evaluation Assessment
Acronym: PANACEA
Status: Active, not recruiting | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Martin Harazim, Dr., Brno University Hospital
Other Study IDs: BrnoUH2024
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Pancreatic Fluid Collection; Acute Pancreatitis
Keywords: acute pancreatis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meropenem Group: Patients with WOPN receiving intravenous meropenem. Serial blood and pancreatic fluid samples were collected to assess drug penetration and pharmacokinetics as part of therapeutic drug monitoring (TDM).
- Piperacillin Group: Patients with WOPN receiving intravenous piperacillin-tazobactam. Serial blood and pancreatic fluid samples were collected to evaluate drug penetration and pharmacokinetics as part of therapeutic drug monitoring (TDM).

SUMMARY:
This observational study aims to evaluate the penetration of intravenously administered antibiotics into pancreatic fluid collections in patients with suspected infected walled-off pancreatic necrosis (WOPN). In selected patients undergoing percutaneous or endoscopic drainage of the collection as part of their clinical care, a small sample of pancreatic fluid will be collected and analyzed to determine the concentration of the administered antibiotic.

At the same time, a blood sample will be taken to assess the antibiotic concentration in plasma. By comparing the concentrations in pancreatic fluid and plasma, the study seeks to determine the extent to which different antibiotics (e.g., meropenem or piperacillin-tazobactam) reach the site of infection within the pancreas.

All procedures performed as part of the study, with the exception of the antibiotic concentration measurement, are standard components of routine care for patients with complicated acute pancreatitis. Participation in the study does not alter the diagnostic or therapeutic management of the patient. Patients provide written informed consent before enrollment.

The results of this study may help optimize antibiotic dosing in patients with infected pancreatic collections and contribute to more effective and individualized treatment strategies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent
* Undergoing percutaneous or endoscopic drainage/puncture of a pancreatic fluid collection

Exclusion Criteria:

- Failure or refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized with past or ongoing acute pancreatitis undergoing drainage or puncture of suspected infected pancreatic fluid collection. Patients are recruited from the University Hospital Brno. Approximately 40 participants are expected.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Antibiotic concentration ratio between pancreatic fluid and plasma | Within 6 hours after antibiotic administration
  Ratio of antibiotic concentration in pancreatic fluid (WOPN) to plasma concentration, determined from simultaneously collected samples after intravenous antibiotic administration

SECONDARY OUTCOMES:
Measured concentrations of antibiotics in pancreatic fluid and plasma | Within 6 hours after antibiotic administration
  Absolute concentrations of meropenem and piperacillin in pancreatic fluid and plasma from simultaneously collected samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Fakultni nemocnice Brno, Brno, Czech Republic, Czechia